CLINICAL TRIAL: NCT03958448
Title: Comparison of Extra-short (4 mm) Implants Used as Distal Support of a Maxillary Full-arch Fixed Dental Prosthesis vs. 10 mm Implants Installed After Sinus Floor Elevation. A Randomized Clinical Trial
Brief Title: Comparison of Extra-short (4 mm) Implants Used as Distal Support of a Maxillary Full-arch Fixed Dental Prosthesis vs. 10 mm Implants Installed After Sinus Floor Elevation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARDEC Academy (Network)
Collaborators: University of Bologna (Other); ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: protocol #15052
Record Dates: First submitted 2019-05-15; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Two groups will be randomly prepared. The Short group, one 4 mm long and 4.1 mm in diameter implant (Short implant) will be installed in each side of the posterior region of the maxilla. The standard group, bilateral sinus floor elevations will be performed. After 4 months of healing, one 10 mm long and 4.1 mm in diameter implant (Standard implant) will be installed into each augmented sinus.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: A statistician not involved in the study performed the randomization in blocks of four and the assignments have been sealed in coded and opaque envelopes that will be opened at the time of the enrollment of each patient in the study. The surgeon will be blinded about the assignment until the time of the surgery. The outcome assessor will be blinded about the protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Group (Experimental): In each side of the posterior region of the maxilla, one tissue level implant, 4 mm long and 4.1 mm in diameter, will be installed
  Interventions: Procedure: Placement of extra short implants
- Standard group (Experimental): sinus floor elevation with will be performed using natural bovine bone graft as filler material and porcine dermis collagen membrane to cover the antrostomy. After 4 months of healing, one bone level implant, 10 mm long and 4.1 mm in diameter, will be installed into each augmented sinus.
  Interventions: Procedure: maxillary sinus lift, maxillary sinus elevation, maxillary sinus augmentation; Procedure: placement of standard implant

INTERVENTIONS:
Procedure: Placement of extra short implants — placement of an extra short implant in the posterior edentulous ridge
  Arms: Short Group
Procedure: maxillary sinus lift, maxillary sinus elevation, maxillary sinus augmentation
  Arms: Standard group
Procedure: placement of standard implant — placement of standard implant in the posterior edentulous ridge after maxillary sinus augmentation
  Arms: Standard group

SUMMARY:
Recently, 4 mm long implants with a standard diameter have been used for the restoration of the posterior edentulous mandible with favorable results. However, randomized clinical trials reporting the results from full-arch fixed dental prosthesis that included 4 mm long implants placed in the posterior regions of the maxilla have not been published yet. The aim of the present study will be to compare the survival and success rates of 4 mm implants used as distal support of a maxillary full-arch fixed dental prosthesis with standard (10 mm) implants placed in association with a bilateral sinus floor augmentation procedure

DETAILED DESCRIPTION:
Two groups will be randomly prepared, the Short group and the Standard group. In the Short group, one 4 mm long and 4.1 mm in diameter implant (extra-short implant) will be installed in each side of the posterior region of the maxilla. In the Standard group, bilateral sinus floor elevations will be performed. After 4 months of healing, one 10 mm long and 4.1 mm in diameter implant (standard implant) will be installed into each augmented sinus. In the frontal region, four 10 mm long implants will be installed in both groups. Clinical assessments and x-rays will be taken at prosthesis delivering (6-8 weeks after implant installation), and after 6, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous maxilla
* Willing to receive a full arch fixed restoration in the maxilla.
* Latest extraction at least 8 weeks before implant insertion
* Sinus floor height included between 4 to 6 mm
* Bone width in the distal segments sufficient to allow the insertion of a 4 mm long implant of standard diameter.
* In the anterior maxilla (from first premolar to first premolar) bone width sufficient to allow the insertion of 10 mm long implants of standard diameter. Minor horizontal augmentations with guided bone regeneration procedures was allowed in the anterior maxilla.

the opposing arch have to present one of the following conditions:

* natural dentition (at least 10 elements from 3.5 to 4.5)
* Fixed dental prosthesis of at least 10 elements (from 3.5 to 4.5) supported by teeth or implants
* Implant supported or teeth supported overdentures
* Adequate partial removable prostheses.

Exclusion Criteria:

* Presence of conditions requiring prophylactic use of antibiotics (e.g., history of rheumatic heart disease, bacterial endocarditis, cardiac valvular anomalies, prosthetic joint replacements).
* Major systemic diseases, or medical conditions requiring prolonged use of steroids, or alcoholism or chronically drug abuse.
* Current pregnancy or breastfeeding women
* Smokers > 10 cigarettes per day
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Immunocompromised patients including patients infected with HIV
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability.
* Patients with an ongoing or previous treatment with bisphosphonates (for at least 2 months for oral therapy or 6 months for IV injection)

Local exclusion criteria

* Local inflammation, including untreated periodontitis
* Pre-cancerous oral lesions
* History of local irradiation therapy
* Severe bruxism or clenching habits
* Patients with inadequate oral hygiene or unmotivated for adequate oral home care
* Previous Guided bone regeneration or Guided tissue regeneration treatment at the implant site
* Total removable prosthesis in the lower arch

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity
Enrollment: 20 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
survival rate of 4 mm implants used as distal support | 24 months
  To compare the survival rates of 4 mm implants used as distal support of a maxillary full-arch fixed dental prosthesis with standard (10 mm) implants placed in association with a bilateral sinus floor augmentation procedure.
Crestal bone level | 24 months
  Change of crestal bone level measured on intraoral x-ray applying a parallel technique from baseline (definitive prosthesis delivering) and 2-year follow-up. The distance between the implant margin and the first bone to implant contact will be measured in millimeters at the mesial and distal aspects of the Short and Standard implants.

SECONDARY OUTCOMES:
Technical complications | 24 months
  Any technical complications related to implants, abutments, screw loosening, prosthetic fracture or chipping of the veneer material expressed in number of occurrence.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pjetursson BE, Tan WC, Zwahlen M, Lang NP. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. J Clin Periodontol. 2008 Sep;35(8 Suppl):216-40. doi: 10.1111/j.1600-051X.2008.01272.x. PMID 18724852
- [Result] Barone A, Ricci M, Grassi RF, Nannmark U, Quaranta A, Covani U. A 6-month histological analysis on maxillary sinus augmentation with and without use of collagen membranes over the osteotomy window: randomized clinical trial. Clin Oral Implants Res. 2013 Jan;24(1):1-6. doi: 10.1111/j.1600-0501.2011.02340.x. Epub 2011 Dec 12. PMID 22151577
- [Result] Masuda K, Silva ER, Botticelli D, Apaza Alccayhuaman KA, Xavier SP. Antrostomy Preparation for Maxillary Sinus Floor Augmentation Using Drills or a Sonic Instrument: A Microcomputed Tomography and Histomorphometric Study in Rabbits. Int J Oral Maxillofac Implants. 2019 July/August;34(4):819-827. doi: 10.11607/jomi.7350. Epub 2019 Feb 15. PMID 30768660
- [Result] Lundgren S, Andersson S, Gualini F, Sennerby L. Bone reformation with sinus membrane elevation: a new surgical technique for maxillary sinus floor augmentation. Clin Implant Dent Relat Res. 2004;6(3):165-73. PMID 15726851
- [Result] Cricchio G, Sennerby L, Lundgren S. Sinus bone formation and implant survival after sinus membrane elevation and implant placement: a 1- to 6-year follow-up study. Clin Oral Implants Res. 2011 Oct;22(10):1200-1212. doi: 10.1111/j.1600-0501.2010.02096.x. PMID 21906186
- [Result] Moon YS, Sohn DS, Moon JW, Lee JH, Park IS, Lee JK. Comparative histomorphometric analysis of maxillary sinus augmentation with absorbable collagen membrane and osteoinductive replaceable bony window in rabbits. Implant Dent. 2014 Feb;23(1):29-36. doi: 10.1097/ID.0000000000000031. PMID 24445918
- [Result] Omori Y, Ricardo Silva E, Botticelli D, Apaza Alccayhuaman KA, Lang NP, Xavier SP. Reposition of the bone plate over the antrostomy in maxillary sinus augmentation: A histomorphometric study in rabbits. Clin Oral Implants Res. 2018 Aug;29(8):821-834. doi: 10.1111/clr.13292. Epub 2018 Jun 7. PMID 29876969
- [Result] Corbella S, Taschieri S, Weinstein R, Del Fabbro M. Histomorphometric outcomes after lateral sinus floor elevation procedure: a systematic review of the literature and meta-analysis. Clin Oral Implants Res. 2016 Sep;27(9):1106-22. doi: 10.1111/clr.12702. Epub 2015 Oct 10. PMID 26452326
- [Result] Caneva M, Lang NP, Garcia Rangel IJ, Ferreira S, Caneva M, De Santis E, Botticelli D. Sinus mucosa elevation using Bio-Oss(R) or Gingistat(R) collagen sponge: an experimental study in rabbits. Clin Oral Implants Res. 2017 Jul;28(7):e21-e30. doi: 10.1111/clr.12850. Epub 2016 Apr 15. PMID 27080163
- [Result] De Santis E, Lang NP, Ferreira S, Rangel Garcia I Jr, Caneva M, Botticelli D. Healing at implants installed concurrently to maxillary sinus floor elevation with Bio-Oss(R) or autologous bone grafts. A histo-morphometric study in rabbits. Clin Oral Implants Res. 2017 May;28(5):503-511. doi: 10.1111/clr.12825. Epub 2016 Mar 10. PMID 26969193
- [Result] Riachi F, Naaman N, Tabarani C, Aboelsaad N, Aboushelib MN, Berberi A, Salameh Z. Influence of material properties on rate of resorption of two bone graft materials after sinus lift using radiographic assessment. Int J Dent. 2012;2012:737262. doi: 10.1155/2012/737262. Epub 2012 Jul 31. PMID 22899930
- [Result] Shanbhag S, Shanbhag V, Stavropoulos A. Volume changes of maxillary sinus augmentations over time: a systematic review. Int J Oral Maxillofac Implants. 2014 Jul-Aug;29(4):881-92. doi: 10.11607/jomi.3472. PMID 25032768
- [Result] Zijderveld SA, van den Bergh JP, Schulten EA, ten Bruggenkate CM. Anatomical and surgical findings and complications in 100 consecutive maxillary sinus floor elevation procedures. J Oral Maxillofac Surg. 2008 Jul;66(7):1426-38. doi: 10.1016/j.joms.2008.01.027. PMID 18571027

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT03958448/Prot_SAP_000.pdf